CLINICAL TRIAL: NCT00379223
Title: Multicenter Trial to Investigate the Safety and Efficacy of Vitrectomy With Radial Optic Neurotomy for the Preservation of Visual Function in Subjects With Central Retinal Vein Occlusion (CRVO)
Brief Title: Radial Optic Neurotomy in Central Retinal Vein Occlusion : a Randomized Trial
Acronym: OVCR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean Pierre LEROY/Clinical Research and innovation Director, University Hospital Bordeaux
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9418-04; 2004-028
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2008-08

CONDITIONS: Retinal Vein Occlusion
Keywords: retinal vein occlusion; vitrectomy; surgery; retinal disorders; vascular diseases
MeSH Terms: conditions — Retinal Vein Occlusion; Retinal Diseases; Vascular Diseases | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Standard treatment of central retinal vein occlusion : the rheologic correction
- 2 (Experimental): Standard treatment of central retinal vein occlusion : the rheologic correction and surgery associating pars plana vitrectomy and radial optic neurotomy
  Interventions: Procedure: vitrectomy with radial optic neurotomy

INTERVENTIONS:
Procedure: vitrectomy with radial optic neurotomy
  Arms: 2

SUMMARY:
Natural evolution of severe central retinal vein occlusion with low visual acuity is very poor. A randomized clinical trial will compare troxerutin and platelet anti-aggregating agents (drug treatment) versus surgery and drug treatment. Surgery will include vitrectomy and radial optic neurotomy. The primary outcome will be vision measured 6 months after surgery.

DETAILED DESCRIPTION:
Central Retinal Vein Occlusion (CRVO) is the second most frequently retinal vascular disease causing loss of vision, after diabetic retinopathy. No treatment of CRVO has clearly demonstrated beneficial and long lasting visual results. Commonly used treatment options are platelet anti-aggregating agents, correcting rheologic factors with troxerutin and isovolumic hemodilution. Surgical treatment of CRVO has recently been proposed (2001) and has been studied in numerous non comparative pilot studies. Limited but encouraging results motivate our randomised controlled trial. We will evaluate at 6 months visual acuity after surgery associating pars plana vitrectomy and radial optic neurotomy, in patients with central vein occlusion and bad vision, associated with the correction of rheologic factors.

ELIGIBILITY:
Inclusion Criteria:

* Central Retinal Vein Occlusion oedematous or hemorrhagic (at fundus exam and at fluorescein angiography)
* Visual Acuity (VA) ≤ 20/200 with ETDRS charts
* Decreased VA since more than 1 month, less than 3 months
* Common care recommendations for CRVO during the period before recruitment (Control ocular pressure if associated hypertension or glaucoma ; Hemodilution if hematocrit ≥ 38% ,if no cardio-vascular contra-indication, to maintain hematocrit under 38% during 6 weeks ; Troxerutin (3 /d) and aspirin (100 - 160 mg/d) ; Clinical and angiographic controls to look for retinal ischemia indicating laser PRP to prevent neovascular glaucoma.
* Signed informed consent.

Exclusion Criteria:

* Ischemic CRVO : 1- More than 30 disc diameters of ischemia at fluorescein angiography and/or •2- If Angiogram is uninterpretable because of hemorrhages, deficit of afferent pupillary reflex 0.9 with photographic filters (proposed by Hayreh) with indication to do laser PRP or laser PRP already done,
* Rubeosis or neovascular glaucoma,
* Bilateral diabetic retinopathy preproliferative or proliferative,
* Uncharacterized coagulation disease, or anticoagulant treatment,
* Untreated systemic disease (diabetes, severe high blood pressure, Cardiac failure) ou eye disease (glaucoma),
* Contra-indication or documented allergy to troxerutin or platelet anti-aggregating agents,
* Contra-indication to surgical procedure
* incapacity to received an informed consent, incapacity to follow all the study schedule

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients showing an improvement of visual acuity (at least 3 lines (15 letters) in ETDRS charts) | between pre operative examination and 6 months after randomization

SECONDARY OUTCOMES:
Efficacy | between pre operative examination and 6 months after randomization
Mean visual acuity | between pre operative examination and 6 months
Macular thickness in Optical Coherence Tomography (OCT)
Persistence of hemorrhages in the fundus
Retinal ischemia indicating pan retinal photocoagulation | 6 months after randomization
Safety : Serious complications after surgery (retinal detachment, retinal ischemia, neovascular glaucoma) or medical treatment during the 6 months following surgery. | after surgery or medical treatment examination and 6 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jean François KOROBELNIK, Pr, Principal Investigator — University Hospital, Bordeaux; Geneviève CHENE, pR, Study Chair — University Hospital, Bordeaux
Locations (1):
- Service d'ophtalmologie, Hopital Pellegrin, place Amélie Raba Léon, Bordeaux, France